CLINICAL TRIAL: NCT05151445
Title: The Use of a Consumer-Based mHealth Dietary App and Health Coaching With Kidney Transplant Recipients
Acronym: TASK
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Tara O'Brien, Assistant Professor at Center for Healthy Aging, Self-Management and Complex Care, Distinguished Educator in Gerontological Nursing/National Hartford Centers of Gerontological Nursing Excellence, Ohio State University
Other Study IDs: 2020B0261
Record Dates: First submitted 2021-11-09; First posted 2021-12-09 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplant; Kidney Transplant; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mHealth dietary app + health coaching intervention: A feasibility study will be utilized to establish the recruitment, retention, and adherence with post-kidney transplant recipients using a consumer-based mHealth dietary app + health coaching.
  Interventions: Behavioral: mHealth dietary app + health coaching intervention

INTERVENTIONS:
Behavioral: mHealth dietary app + health coaching intervention — The "Lose-It" app will be set up with Gmail accounts with unique unidentifiable codes developed by the research team. Participants be trained to enter their dietary intake and physical activity daily for 12-weeks. Participants will monitor their vegetable intake, fat intake, carbohydrate intake, weight, and blood pressure. Wi-Fi connected weight scales and blood pressure cuff will be supplied for weight and blood pressure monitoring. Participants will be taught how to sync the data from the scales and blood pressure cuff to the app for the research team to access. Participants will perform a return demonstration to confirm that they can record their dietary intake daily, physical activity, weight, and blood pressure using the "Lose-It" app. We also review with the participant the "My Plate" method for proper nutrition and the steps to distance conversion chart.

SUMMARY:
The purpose of the study is to test the feasibility mHealth dietary app + health coaching for improving primary outcomes (recruitment, retention, and adherence) and secondary outcomes (perceived stress [ Perceived Stress Scale], exercise self-efficacy[Exercise Self-efficacy Scale], vegetable intake [Fruit, Vegetables, and Fiber Screen] fat intake [Lose-it Premium database], carbohydrate intake [Lose-it Premium database], weight, [Wi-Fi weight scale using the Lose-it Premium database], and blood pressure [Wi-Fi blood pressure cuff using the Lose-it Premium database].

DETAILED DESCRIPTION:
The proposed study seeks to shift the paradigm for promoting diet intake and physical activity using education and self-report to provide a powerful combination of mHealth dietary app and health coaching (set goals, provide ongoing feedback, and self-monitor behaviors). To the investigators knowledge, this is the first time a mHealth dietary app and health coaching intervention has been used in kidney transplant recipients to link real-time data for monitoring dietary intake and physical activity.

The long-term goal of this work is to enhance well-being in kidney recipients via lifestyle self-management of care for dietary intake and physical activity to ultimately prevent chronic diseases. The proposed study is important because early weight gain after kidney transplant is associated with adverse effects on the transplanted kidney function resulting in increased health care cost and poor quality of life. Interventions are needed to monitor kidney transplant recipients diet and physical activity in real-time to prevent health decline.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older men and women
* functioning KTR (not on dialysis)
* ability to speak, read, and hear English,
* possession of a smartphone capable of accessing and downloading a mHealth dietary app
* Wi-Fi or Internet access,
* greater than 3 months post-transplant (due to medication adjustments and decreased functional levels),
* not hospitalized
* capable of self-consent per capacity screening.

Exclusion Criteria:

* Participation in a weight loss program
* participation in a structured exercise program
* diagnosis of dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited or contacted from a list of kidney recipients that have already requested they be contacted for future studies from our previous study. This list consists of approximately 60 people.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conte C, Secchi A. Post-transplantation diabetes in kidney transplant recipients: an update on management and prevention. Acta Diabetol. 2018 Aug;55(8):763-779. doi: 10.1007/s00592-018-1137-8. Epub 2018 Apr 4. PMID 29619563
- [Background] Aksoy N. Weight Gain After Kidney Transplant. Exp Clin Transplant. 2016 Nov;14(Suppl 3):138-140. PMID 27805534
- [Background] Zelle DM, Kok T, Dontje ML, Danchell EI, Navis G, van Son WJ, Bakker SJ, Corpeleijn E. The role of diet and physical activity in post-transplant weight gain after renal transplantation. Clin Transplant. 2013 Jul-Aug;27(4):E484-90. doi: 10.1111/ctr.12149. Epub 2013 Jun 13. PMID 23758229
- [Background] Workeneh B, Moore LW, Nolte Fong JV, Shypailo R, Gaber AO, Mitch WE. Successful Kidney Transplantation Is Associated With Weight Gain From Truncal Obesity and Insulin Resistance. J Ren Nutr. 2019 Nov;29(6):548-555. doi: 10.1053/j.jrn.2019.01.009. Epub 2019 Mar 7. PMID 30852120
- [Background] Rosenberger J, Geckova AM, Dijk JP, Roland R, Heuvel WJ, Groothof F JW. Factors modifying stress from adverse effects of immunosuppressive medication in kidney transplant recipients. Clin Transplant. 2005 Feb;19(1):70-6. doi: 10.1111/j.1399-0012.2004.00300.x. PMID 15659137
- [Background] Klaassen G, Zelle DM, Navis GJ, Dijkema D, Bemelman FJ, Bakker SJL, Corpeleijn E. Lifestyle intervention to improve quality of life and prevent weight gain after renal transplantation: Design of the Active Care after Transplantation (ACT) randomized controlled trial. BMC Nephrol. 2017 Sep 15;18(1):296. doi: 10.1186/s12882-017-0709-0. PMID 28915863
- [Background] Kim IK, Choi SH, Son S, Ju MK. Early Weight Gain After Transplantation Can Cause Adverse Effect on Transplant Kidney Function. Transplant Proc. 2016 Apr;48(3):893-6. doi: 10.1016/j.transproceed.2015.10.064. PMID 27234761
- [Background] Edwards ES, Sackett SC. Psychosocial Variables Related to Why Women are Less Active than Men and Related Health Implications. Clin Med Insights Womens Health. 2016 Jul 4;9(Suppl 1):47-56. doi: 10.4137/CMWH.S34668. eCollection 2016. PMID 27398045
- [Background] Hap K, Madziarska K, Hap W, Zmonarski S, Zielinska D, Kaminska D, Banasik M, Koscielska-Kasprzak K, Klinger M, Mazanowska O. Are Females More Prone Than Males to Become Obese After Kidney Transplantation? Ann Transplant. 2019 Jan 29;24:57-61. doi: 10.12659/AOT.912096. PMID 30737367
- [Background] Pedrollo EF, Nicoletto BB, Carpes LS, de Freitas JMC, Buboltz JR, Forte CC, Bauer AC, Manfro RC, Souza GC, Leitao CB. Effect of an intensive nutrition intervention of a high protein and low glycemic-index diet on weight of kidney transplant recipients: study protocol for a randomized clinical trial. Trials. 2017 Sep 6;18(1):413. doi: 10.1186/s13063-017-2158-2. PMID 28874181
- [Background] Wilcox J, Waite C, Tomlinson L, Driscoll J, Karim A, Day E, Sharif A. Comparing glycaemic benefits of Active Versus passive lifestyle Intervention in kidney Allograft Recipients (CAVIAR): study protocol for a randomised controlled trial. Trials. 2016 Aug 22;17(1):417. doi: 10.1186/s13063-016-1543-6. PMID 27550305
- [Background] Clunk JM, Lin CY, Curtis JJ. Variables affecting weight gain in renal transplant recipients. Am J Kidney Dis. 2001 Aug;38(2):349-53. doi: 10.1053/ajkd.2001.26100. PMID 11479161
- [Background] Aminu MS, Sagren N, Manga P, Nazir MS, Naicker S. Obesity and graft dysfunction among kidney transplant recipients: Increased risk for atherosclerosis. Indian J Nephrol. 2015 Nov-Dec;25(6):340-3. doi: 10.4103/0971-4065.151358. PMID 26664208
- [Background] Williams-Hooker R, Draper CM, Chen L, Mitchell CO, Cashion AK. The relationship between fruit and vegetable consumption and weight gain in kidney transplant recipients within 1 year posttransplant. Top Clin Nutr. 2015;30(4):324-332.
- [Background] Mellen PB, Gao SK, Vitolins MZ, Goff DC Jr. Deteriorating dietary habits among adults with hypertension: DASH dietary accordance, NHANES 1988-1994 and 1999-2004. Arch Intern Med. 2008 Feb 11;168(3):308-14. doi: 10.1001/archinternmed.2007.119. PMID 18268173
- [Background] Zeltzer SM, Taylor DO, Tang WH. Long-term dietary habits and interventions in solid-organ transplantation. J Heart Lung Transplant. 2015 Nov;34(11):1357-65. doi: 10.1016/j.healun.2015.06.014. Epub 2015 Jul 6. PMID 26250965
- [Background] O'Brien T, Jenkins C, Amella E, Mueller M, Moore M, Hathaway D. An Internet-Assisted Weight Loss Intervention for Older Overweight and Obese Rural Women: A Feasibility Study. Comput Inform Nurs. 2016 Nov;34(11):513-519. doi: 10.1097/CIN.0000000000000275. PMID 27392256
- [Background] Boehmer KR, Barakat S, Ahn S, Prokop LJ, Erwin PJ, Murad MH. Health coaching interventions for persons with chronic conditions: a systematic review and meta-analysis protocol. Syst Rev. 2016 Sep 1;5(1):146. doi: 10.1186/s13643-016-0316-3. PMID 27585627
- [Background] Wolever RQ, Simmons LA, Sforzo GA, Dill D, Kaye M, Bechard EM, Southard ME, Kennedy M, Vosloo J, Yang N. A Systematic Review of the Literature on Health and Wellness Coaching: Defining a Key Behavioral intervention in Healthcare. Glob Adv Health Med. 2013 Jul;2(4):38-57. doi: 10.7453/gahmj.2013.042. PMID 24416684
- [Background] O'Brien T, Troutman-Jordan M, Hathaway D, Armstrong S, Moore M. Acceptability of wristband activity trackers among community dwelling older adults. Geriatr Nurs. 2015 Mar-Apr;36(2 Suppl):S21-5. doi: 10.1016/j.gerinurse.2015.02.019. Epub 2015 Mar 13. PMID 25771957
- [Background] O'Brien T, Russell CL, Tan A, Mion L, Rose K, Focht B, Daloul R, Hathaway D. A Pilot Randomized Controlled Trial Using SystemCHANGE Approach to Increase Physical Activity in Older Kidney Transplant Recipients. Prog Transplant. 2020 Dec;30(4):306-314. doi: 10.1177/1526924820958148. Epub 2020 Sep 10. PMID 32912051
- [Background] O'Brien T, Hathaway D. An Integrative Literature Review of Physical Activity Recommendations for Adult Renal Transplant Recipients. Prog Transplant. 2016 Dec;26(4):381-385. doi: 10.1177/1526924816664079. Epub 2016 Sep 20. PMID 27555071
- [Background] O'Brien T, Hathaway D, Russell CL, Moore SM. Merging an Activity Tracker with SystemCHANGE to Improve Physical Activity in Older Kidney Transplant Recipients. Nephrol Nurs J. 2017 Mar-Apr;44(2):153-157. PMID 29165966
- [Background] O'Brien T, Russell CL, AlKahlout N, Rosenthal A, Meyer T, Tan A, Daloul R, Hathaway D. Recruitment of Older Kidney Transplant Recipients to a Longitudinal Study. Nurs Res. 2020 May/Jun;69(3):233-237. doi: 10.1097/NNR.0000000000000406. PMID 31688340
- [Background] O'Brien T, Meyer T. A Feasibility Study for Teaching Older Kidney Transplant Recipients How to Wear and Use an Activity Tracker to Promote Daily Physical Activity. Nephrol Nurs J. 2020 Jan-Feb;47(1):47-51. PMID 32083436
- [Background] O'Brien T, Russell CL, Tan A, Washington M, Hathaway D. An Exploratory Correlational Study in the Use of Mobile Technology Among Adult Kidney Transplant Recipients. Prog Transplant. 2018 Dec;28(4):368-375. doi: 10.1177/1526924818800051. Epub 2018 Sep 24. PMID 30249156
- [Background] Moore SM, Jones L, Alemi F. Family self-tailoring: Applying a systems approach to improving family healthy living behaviors. Nurs Outlook. 2016 Jul-Aug;64(4):306-311. doi: 10.1016/j.outlook.2016.05.006. Epub 2016 May 18. PMID 27301950
- [Background] Deming WE, Orsini JN. The essential Deming : leadership principles from the father of quality management. New York: McGraw-Hill; 2013.
- [Background] Resnick B, Gruber-Baldini AL, Pretzer-Aboff I, Galik E, Buie VC, Russ K, Zimmerman S. Reliability and validity of the evaluation to sign consent measure. Gerontologist. 2007 Feb;47(1):69-77. doi: 10.1093/geront/47.1.69. PMID 17327542
- [Background] Sundararajan V, Quan H, Halfon P, Fushimi K, Luthi JC, Burnand B, Ghali WA; International Methodology Consortium for Coded Health Information (IMECCHI). Cross-national comparative performance of three versions of the ICD-10 Charlson index. Med Care. 2007 Dec;45(12):1210-5. doi: 10.1097/MLR.0b013e3181484347. PMID 18007172
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Sun Y, Gao L, Kan Y, Shi BX. The Perceived Stress Scale-10 (PSS-10) is reliable and has construct validity in Chinese patients with systemic lupus erythematosus. Lupus. 2019 Feb;28(2):149-155. doi: 10.1177/0961203318815595. Epub 2018 Dec 5. PMID 30518288
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Block G, Gillespie C, Rosenbaum EH, Jenson C. A rapid food screener to assess fat and fruit and vegetable intake. Am J Prev Med. 2000 May;18(4):284-8. doi: 10.1016/s0749-3797(00)00119-7. PMID 10788730
- [Derived] O'Brien T, Rose K, Focht B, Al Kahlout N, Jensen T, Heareth K, Nori U, Daloul R. The feasibility of Technology, Application, Self-Management for Kidney (TASK) intervention in post-kidney transplant recipients using a pre/posttest design. Pilot Feasibility Stud. 2023 Nov 22;9(1):190. doi: 10.1186/s40814-023-01417-9. PMID 37993961
- See also: National Institute of Diabetes and Digestive and Kidney Diseases. Mission & Vision. 2019 Accessed August, 30, 2019 — http://www.niddk.nih.gov/about-niddk/meet-director/mission-vision

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of of participatns took place among patients who received care at a Midwest Medical Center Kidney Transplant Clinic or attended a Midwest transplant support group over four months using a convenience sampling strategy. Eligibility criteria for this study consisted of KRs, age 18 years or older, not on dialysis, the ability to speak and hear English, and possession of a smartphone capable of accessing and downloading mobile applications (apps), Wi-Fi, or Internet access.
Pre-assignment Details: Participants were not eligible for this study if they were participating in a weight loss or structured exercise program or could not pass a brief cognitive test.
Period: Overall Study
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Started (Intended recruitment goal for study was 20) | 20
Week 4 | 18
Week 8 | 18
Completed | 17
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.45 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Employment [Count of Participants; unit: Participants]
  Full-time employment | 5
  Not employed | 9
  Retired | 6
Number of kidney transplants [Count of Participants; unit: Participants]
  1 | 18
  2 + | 2
Type of transplant [Count of Participants; unit: Participants]
  Deceased donor | 14
  Living donor | 6
Caregiver [Count of Participants; unit: Participants]
  Self | 18
  Spouse or partner | 1
  Parent or legal guardian | 1
Number of household members [Count of Participants; unit: Participants]
  1 | 3
  2 | 11
  3 | 4
  4 | 2
Income [Count of Participants; unit: Participants]
  Under $20,000 | 1
  $20,000-$45,000 | 5
  $46,000-$65,000 | 5
  $91,000-$125,000 | 6
  $126,000 + | 3
Education [Count of Participants; unit: Participants]
  High School Diploma or GED | 4
  Associate's or Technical | 5
  Bachelor's | 7
  Master's | 4

OUTCOME MEASURES:

1. Primary Outcome: The Feasibility of the Study Recruitment for the Study
Description: Recruitment (percent of participants approached to be in the study), will be recorded by the research assistant.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: The Feasibility of Participant Retention for the Study
Description: Retention (percent of participants that dropped during the study), will be recorded by the research assistant.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
Participants
  Baseline | 20
  4 weeks | 18
  8 weeks | 18
  12 weeks | 17

3. Primary Outcome: The Feasibility of Adherence for Using the Lose- It App to Record Diet
Description: Adherence (percent to adhere to logging daily dietary intake) will be recorded continuously each day by the "Lose-It" app.
Time Frame: Weekly for 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 18
Participants
  Week 1 | 17
  Week 2 | 17
  Week 3 | 17
  Week 4 | 16
  Week 5 | 16
  Week 6 | 16
  Week 7 | 15
  Week 8 | 16
  Week 9 | 17
  Week 10 | 16
  Week 11 | 15
  Week 12 | 15

4. Primary Outcome: The Feasibility of Adherence for Using the Lose- It App to Physical Actvity
Description: Adherence (percent to adhere to logging daily physical activity) will be recorded continuously each day by the "Lose-It" app.
Time Frame: Weekly for 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 18
Participants
  Week 1 | 5
  Week 2 | 5
  Week 3 | 6
  Week 4 | 5
  Week 5 | 3
  Week 6 | 3
  Week 7 | 5
  Week 8 | 4
  Week 9 | 6
  Week 10 | 5
  Week 11 | 5
  Week 12 | 3

5. Secondary Outcome: Perceived Stress Level
Description: Perceived Stress Scale will be evaluated by using the Perceived Stress Scale (PSS).The PSS is a 10-item questionnaire using a Likert Scale to rate feelings of stress from 0 "never" to 4 "very often." Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Population: There were some participants who withdrew from the study over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
score on a scale
  Baseline | 21.65 (3.88)
  Week 4: number analyzed (Participants) | 18
  Week 4 | 17.56 (5.03)
  Week 8: number analyzed (Participants) | 18
  Week 8 | 18.00 (4.79)
  Week 12: number analyzed (Participants) | 17
  Week 12 | 18.82 (5.27)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.002, McNemar; 95% CI = -3.56, 95% CI 2-sided [-5.65 to -1.46]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.004, McNemar; 95% CI = -3.11, 95% CI 2-sided [-5.07 to -1.15]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.038, McNemar; 95% CI = -2.53, 95% CI 2-sided [-4.90 to 0.16]

6. Secondary Outcome: Exercise Self-Efficacy
Description: Exercise Self-Efficacy Scale will be evaluated by using the Self-Efficacy for Exercise (SEE) Scale. The SEE is a 9-item questionnaire using a Likert Scale to rate feelings of stress from 0 "not confident" to 10 "very confident." This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
score on a scale
  Baseline | 60.75 (23.35)
  Week 4 | 71.00 (18.69)
  Week 8 | 71.17 (17.67)
  Week 12 | 80.71 (17.68)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.062, McNemar; 95% CI = 9.61, 95% CI 2-sided [-0.55 to 19.77]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.098, McNemar; 95% CI = 9.78, 95% CI 2-sided [-2.01 to 21.56]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.003, McNemar; 95% CI = 17.06, 95% CI 2-sided [6.51 to 27.60]

7. Secondary Outcome: Fruit and Vegetable Servings Per Day
Description: Fruit and vegetable intake will be assessed using the Fruit, Vegetable and Fiber Screen which uses a scale to assess fruit and vegetable intake using a Likert Scale to rate intake from less than1/ per week to more than 2 a day. Higher scores indicate that more fruits and vegetables are being consumed by participants.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Number; unit: servings of fruit and vegetables per day
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
servings of fruit and vegetables per day
  Baseline - 2 Servings or Less | 11
  Basline - 3 Servings or More | 8
  Week 4 - 2 Servings or Less | 8
  Week 4 - 3 Servings or More | 10
  Week 8 - 2 Servings or Less | 9
  Week 8 - 3 Servings or More | 9
  Week 12 - 2 Servings or Less | 7
  Week 12 - 3 Servings or More | 10
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.37, McNemar
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.724, McNemar
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.289, McNemar

8. Secondary Outcome: Fiber Intake
Description: Fiber intake will be assessed using the Fruit, Vegetable and Fiber Screen which uses a scale to assessfiber intake using a Likert Scale to rate intake from less than1/ per week to more than 2 a day.Higher scores indicate more fiber intake.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
Participants
  Baseline - 20 mg or Less | 16
  Baseline - 21 mg or More | 3
  Week 4 - 20 mg or Less | 15
  Week 4 - 21 mg or More | 3
  Week 8 - 20 mg or Less | 15
  Week 8 - 21 mg or More | 3
  Week 12 - 20 mg or Less | 14
  Week 12 - 21 mg or More | 4
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 1.000, McNemar
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 1.000, McNemar
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Weel 12 vs. Baseline; Test type: Other; p = 1.000, McNemar

9. Secondary Outcome: Fat Intake
Description: The participant will record their percent of fat intake each day into the Lose-it Premium application.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of fat intake
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
percentage of fat intake
  Baseline | 29.59 (14.17)
  Week 4 | 28.49 (9.07)
  Week 8 | 28.51 (7.59)
  Week 12 | 25.98 (6.44)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.696, McNemar; 95% CI = -1.1, 95% CI 2-sided [-6.96 to 4.76]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.734, McNemar; 95% CI = -1.08, 95% CI 2-sided [-7.72 to 5.56]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.249, McNemar; 95% CI = -4.15, 95% CI 2-sided [-11.53 to 3.23]

10. Secondary Outcome: Carbohydrate Intake
Description: The participant will record their percent of carbohydrate intake each day into the Lose-it Premium application.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of carbohydrate intake
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
percentage of carbohydrate intake
  Baseline | 32.69 (9.42)
  Week 4 | 32.65 (8.76)
  Week 8 | 36.12 (11.11)
  Week 12 | 33.24 (10.17)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.989, McNemar; 95% CI = -0.04, 95% CI 2-sided [-5.25 to 5.18]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.263, McNemar; 95% CI = 3.43, 95% CI 2-sided [-2.83 to 9.69]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.882, McNemar; Slope = 0.44, 95% CI 2-sided [-5.80 to 6.68]

11. Secondary Outcome: Weight
Description: Weight (pounds) will be measured each day by the participant using a wireless Wi Fi weight scale. The data from the wireless weight scale will sync the data from the participant's mobile phone to the premium password-protect "Lose-It" database each day.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
pounds
  Basline | 190.11 (44.57)
  Week 4 | 189.48 (44.84)
  Week 8 | 182.88 (38.36)
  Week 12 | 186.61 (47.02)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.425, McNemar; 95% CI = -0.62, 95% CI 2-sided [-2.23 to 0.98]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.205, McNemar; 95% CI = -4.98, 95% CI 2-sided [-9.08 to -0.88]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.020, McNemar; 95% CI = -4.98, 95% CI 2-sided [-9.08 to -0.8]

12. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (millimeters of mercury [mmHg]) will be recorded each day by the participant using a wireless Wi Fi blood pressure cuff. The data from the wireless cuff will sync from the participant's mobile phone to the premium password-protect "Lose-It" database each day.
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
millimeters of mercury (mmHg)
  Baseline | 134.28 (27.46)
  Week 4 | 137.33 (20.92)
  Week 8 | 129.89 (26.22)
  Week 12 | 128.47 (18.99)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.429, McNemar; 95% CI = 0.429, 95% CI 2-sided [-4.90 to 11.01]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.255, McNemar; 95% CI = -4.39, 95% CI 2-sided [-12.24 to 3.46]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = 0.102, McNemar; 95% CI = -7.00, 95% CI 2-sided [-15.55 to 1.55]

13. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 12
Time Frame: Assessed at Baseline, 4 weeks, 8 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | mHealth Dietary App + Health Coaching Intervention
Number analyzed (Participants) | 20
millimeters of mercury (mmHg)
  Baseline | 80.39 (16.67)
  Week 4 | 78.44 (10.02)
  Week 8 | 76.28 (11.27)
  Week 12 | 76.94 (11.83)
Statistical Analysis 1: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 4 vs. Baseline; Test type: Other; p = 0.568, McNemar; 95% CI = -1.94, 95% CI 2-sided [-8.99 to 5.10]
Statistical Analysis 2: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 8 vs. Baseline; Test type: Other; p = 0.198, McNemar; 95% CI = -4.11, 95% CI 2-sided [-10.59 to 2.37]
Statistical Analysis 3: Comparison: mHealth Dietary App + Health Coaching Intervention; Week 12 vs. Baseline; Test type: Other; p = .225, McNemar; 95% CI = -3.76, 95% CI 2-sided [-10.08 to 2.55]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | mHealth Dietary App + Health Coaching Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT05151445/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT05151445/ICF_001.pdf